CLINICAL TRIAL: NCT02653625
Title: PERSEUS: A Phase 2 Proof of Concept Study Investigating the Preliminary Efficacy and Safety of Cenicriviroc in Adult Subjects With Primary Sclerosing Cholangitis (PSC)
Brief Title: PERSEUS: Preliminary Efficacy and Safety of Cenicriviroc in Adult Participants With Primary Sclerosing Cholangitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tobira Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 652-205
Record Dates: First submitted 2016-01-08; First posted 2016-01-12 (Estimated); Results first posted 2018-10-01 (Actual); Last update posted 2018-10-01 (Actual); Status verified 2018-08

CONDITIONS: Primary Sclerosing Cholangitis
Keywords: Primary Sclerosing Cholangitis
MeSH Terms: conditions — Cholangitis, Sclerosing | interventions — cenicriviroc

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cenicriviroc 150 mg (Experimental): One tablet of Cenicriviroc 150 mg once daily with food in the morning for 24 weeks.
  Interventions: Drug: Cenicriviroc 150 mg

INTERVENTIONS:
Drug: Cenicriviroc 150 mg — One tablet of CVC 150 mg once daily taken with food in the morning.
  Other Names: CVC 150 mg

SUMMARY:
This is an open label, proof of concept (PoC) study of Cenicriviroc (CVC) in adult participants with Primary Sclerosing Cholangitis (PSC). The main objective of this PoC study is to assess changes in alkaline phosphatase (ALP) both individually and as a group, over 24 weeks of treatment with CVC.

ELIGIBILITY:
Inclusion Criteria:

* Participants with chronic cholestatic liver disease for at least 6 months
* Clinical diagnosis of Primary Sclerosing Cholangitis (PSC) as evident by chronic cholestasis of more than six months duration with either a consistent magnetic resonance cholangiopancreatography (MRCP)/endoscopic retrograde cholangiopancreatography (ERCP) showing sclerosing cholangitis, or a liver biopsy taken at any time consistent with PSC in the absence of a documented alternative etiology for sclerosing cholangitis. If diagnosis of PSC was made by histology alone, it must require the presence of fibro-obliterative lesions (i.e., onion skin lesions)
* Participants with or without Inflammatory Bowel Disease (IBD) are allowed. If participant has IBD, documented evidence of IBD either by prior endoscopy or in previous medical records, for ≥ 6 months. In addition, participants will be required to enter the study with a Partial Mayo Risk score of 0-3, inclusively
* In participants receiving treatment with ursodeoxycholic acid (UDCA), therapy must be stable for at least 3 months, and at a dose not greater than 20 mg/kg/day
* Serum ALP greater than 1.5 × upper limit of normal (ULN)
* Ability to understand and sign a written informed consent form (ICF)
* Participants receiving allowed concomitant medications need to be on stable therapy for 28 days prior to the Baseline Visit with the exception of UDCA in which participants need to be on stable therapy for ≥ 3 months

Exclusion Criteria:

* Presence of documented secondary sclerosing cholangitis (such as ischemic cholangitis, recurrent pancreatitis, intraductal stone disease, severe bacterial cholangitis, surgical or blunt abdominal trauma, recurrent pyogenic cholangitis, choledocholithiasis, toxic sclerosing cholangitis due to chemical agents, or any other cause of secondary sclerosing cholangitis) on prior clinical investigations
* Small duct PSC
* Presence of percutaneous drain or bile duct stent
* History of cholangiocarcinoma or high clinical suspicion over dominant stricture within 1 year by MRCP/ERCP or clinical judgment
* Ascending cholangitis within 60 days prior to Screening
* Alcohol consumption greater than 21 units/week for males or 14 units/week for females (one unit of alcohol is ½ pint of beer [285 mL], 1 glass of spirits [25 mL] or 1 glass of wine [125 mL])
* Prior or planned liver transplantation
* Presence of alternative causes of chronic liver disease, including alcoholic liver disease, non-alcoholic steatohepatitis, primary biliary cirrhosis, autoimmune hepatitis
* History of cirrhosis and/or hepatic impairment (Child-Pugh classes A, B and C) and/or hepatic decompensation including ascites, encephalopathy or variceal bleeding. Participants who show evidence of significant worsening of hepatic function will be excluded
* Participants with fibrosis evidence of cirrhosis, as determined by local transient elastography (TE, e.g., Fibroscan) values of ≥ 13.0 kPa, taken within the last 6 months. If TE has not been conducted within the 6 months prior to screening, then one will be conducted during the screening period and can be used as the Baseline value.
* Moderate to Severe active IBD or flare in colitis activity within the last 90 days requiring intensification of therapy beyond Baseline treatment. Participants with stable mild to moderate IBD, who are on treatment, are allowed provided they are stable for 3 months with 5-amino salicylic acid drugs or Azathioprine (allowed dose of azathioprine is 50-200 mg/day)
* Use of oral prednisolone > 10 mg/day, biologics and/or hospitalization for colitis within 90 days are disallowed
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT); above the allowed cut-offs, as determined by Screening values:

  * AST > 200 IU/L males and females
  * ALT: males > 250 IU/L and females > 200 IU/L
* Total Bilirubin and Direct Bilirubin; above the allowed cut-offs, as determined by Screening values:

  * Total Bilirubin > 2.0 mg/dL
  * Direct Bilirubin > 0.8 mg/dL
* International normalized ratio > 1.3 in the absence of anticoagulants
* Immunoglobulin G4 (IgG4) > 4 × ULN at Screening or evidence of IgG4-related sclerosing cholangitis
* Females who are pregnant or breastfeeding
* Any other clinically significant disorders or prior therapy that, in the opinion of the investigator, would make the participant unsuitable for the study or unable to comply with the dosing and protocol requirements

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-03-14 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J.P. Nicandro, Study Director — Allergan
Locations (9):
- United States (5):
  - Scripps Clinic, La Jolla, California
  - University of California, Davis Medical Center, Sacramento, California
  - Sutter Health, California Pacific Medical Center, San Francisco, California
  - University of Miami, Miami, Florida
  - Icahn School of Medicine, New York, New York
- Canada (4):
  - University of Calgary, Liver Unit, Calgary, Alberta
  - University of Alberta, Zeidler Ledcor Centre, Edmonton, Alberta
  - University of Manitoba, Winnipeg, Manitoba
  - Toronto University Health Center, Toronto, Ontario

REFERENCES:
- [Derived] Eksteen B, Bowlus CL, Montano-Loza AJ, Lefebvre E, Fischer L, Vig P, Martins EB, Ahmad J, Yimam KK, Pockros PJ, Feld JJ, Minuk G, Levy C. Efficacy and Safety of Cenicriviroc in Patients With Primary Sclerosing Cholangitis: PERSEUS Study. Hepatol Commun. 2020 Dec 22;5(3):478-490. doi: 10.1002/hep4.1619. eCollection 2021 Mar. PMID 33681680

RESULTS

PARTICIPANT FLOW:
Groups:
- Cenicriviroc 150 mg: Cenicriviroc 150 mg was administered orally once daily with food in the morning for 24 weeks.
Period: Overall Study
Arm/Group | Cenicriviroc 150 mg
Started | 24
Completed | 20
Not Completed | 4
Not completed — Adverse Event | 1
Not completed — Non-compliance with Study Drug | 1
Not completed — Protocol Violation | 1
Not completed — Suspected Drug Induced Liver Injury | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) and Safety Analysis Sets: All enrolled participants who received at least 1 dose of study treatment.
Arm/Group | Cenicriviroc 150 mg
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.3 (12.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 21
  Black or African American | 1
  Asian | 1
  Other | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 2
  Not Hispanic | 22

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change From Baseline Through Week 24 in Serum Alkaline Phosphatase (ALP)
Description: ALP was used as a primary surrogate marker for measuring Primary Sclerosing Cholangitis disease. The percent change from Baseline was defined as 100*(value at each visit - Baseline value)/Baseline value. The Baseline value was defined as the last non-missing value on or before the Baseline visit (Day 1). A negative percentage change from baseline indicates an improvement.
Time Frame: Baseline (Day 1) to Week 24
Population: ITT Population: All enrolled participants who received at least 1 dose of study treatment. Participants who did not return for any post-baseline visits were not included in the efficacy measurements. Number of participants analyzed are the participants with available data at the given time-point.
Measure: Mean (Standard Deviation); unit: percentage change in ALP
Arm/Group | Cenicriviroc 150 mg
Number analyzed (Participants) | 20
percentage change in ALP | -4.5 (34.84)

2. Secondary Outcome: Percentage of Participants Who Normalized ALP at Week 24
Description: ALP was used as a primary surrogate marker for measuring Primary Sclerosing Cholangitis disease. Normalization was defined as ALP values outside of the central laboratory reference range at baseline, but within the central laboratory reference range at Week 24.
Time Frame: Week 24
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Cenicriviroc 150 mg
Number analyzed (Participants) | 20
percentage of participants | 0.0 [0.83 to 1.00]

3. Secondary Outcome: Percentage of Participants Who Achieved Serum ALP of Less Than 1.5 Times Upper Limit of Normal (ULN) in Serum ALP at Week 24
Description: ALP was used as a primary surrogate marker for measuring Primary Sclerosing Cholangitis disease. The upper limit of normal ALP was defined according to the central laboratory reference ranges.
Time Frame: Week 24
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Cenicriviroc 150 mg
Number analyzed (Participants) | 20
percentage of participants | 10 [0.68 to 0.98]

4. Secondary Outcome: Percentage of Participants Who Achieved a 50% Decrease in ALP at Week 24
Description: ALP was used as a primary surrogate marker for measuring Primary Sclerosing Cholangitis disease.
Time Frame: Week 24
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Cenicriviroc 150 mg
Number analyzed (Participants) | 20
percentage of participants | 0.0 [0.83 to 1.00]

5. Secondary Outcome: Percentage of Participants With a Treatment-emergent Adverse Event (TEAE)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, regardless of whether related to the medicinal (investigational) product. A TEAE was defined as an AE with an onset that occurred after receiving treatment.
Time Frame: Baseline (Day 1) to Week 24
Population: Safety Analysis Set: All enrolled participants who received at least 1 dose of study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Cenicriviroc 150 mg
Number analyzed (Participants) | 24
percentage of participants | 83.3

6. Secondary Outcome: Percentage of Participants Who Discontinued Due to a TEAE
Description: An adverse event was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, regardless of whether related to the medicinal (investigational) product. A TEAE was defined as an AE with an onset that occurred after receiving treatment.
Time Frame: Baseline (Day 1) to Week 24
Population: Safety Analysis Set: All enrolled participants who received at least 1 dose of study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Cenicriviroc 150 mg
Number analyzed (Participants) | 24
percentage of participants | 8.3

ADVERSE EVENTS:
Time Frame: From Baseline (Day 1) to Week 24
Description: Safety Analysis Set: All enrolled participants who received at least 1 dose of study treatment.
Arm/Group | Cenicriviroc 150 mg
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 1/24
Other Adverse Events (participants affected / at risk) | 20/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cenicriviroc 150 mg (N=24)
Gallbladder polyp (Hepatobiliary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cenicriviroc 150 mg (N=24)
Rash (Skin and subcutaneous tissue disorders) | 4
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash pruritic (Skin and subcutaneous tissue disorders) | 2
Vomiting (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 2
Fatigue (General disorders) | 4
Pyrexia (General disorders) | 2
Dizziness (Nervous system disorders) | 4
Headache (Nervous system disorders) | 3
Lower respiratory tract infection (Infections and infestations) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2016-06-14): https://cdn.clinicaltrials.gov/large-docs/25/NCT02653625/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-12): https://cdn.clinicaltrials.gov/large-docs/25/NCT02653625/SAP_001.pdf